CLINICAL TRIAL: NCT05823792
Title: Comparison of Artificial Intelligence and Ultrasonographers With Different Skills in Diagnosing Intussusception in Children and Identifying Indications for Surgery
Brief Title: Performance of Artificial Intelligence Tools and Ultrasonographers With Different Skills
Acronym: PAITUWDS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hongkui Yu， MD (Other)
Responsible Party: Sponsor-Investigator, Hongkui Yu， MD, Chief Physician, Guangzhou Women and Children's Medical Center
Organization: Guangzhou Women and Children's Medical Center (Other)
Other Study IDs: GuangzhouWCMC20230409
Record Dates: First submitted 2023-04-09; First posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Ileocolic Intussusception

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples Without DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients aged 3-36 months with suspected ileocolic intussusception: Patients aged 3-36 months with suspected ileocolic intussusception
  Interventions: Diagnostic Test: Non-invasive diagnosis of ileocolic intussusception by ultrasound with indication for surgery

INTERVENTIONS:
Diagnostic Test: Non-invasive diagnosis of ileocolic intussusception by ultrasound with indication for surgery — Non-invasive diagnosis of ileocolic intussusception by ultrasound with indication for surgery

SUMMARY:
Artificial intelligence versus different skilled sonographers.

DETAILED DESCRIPTION:
Comparison of artificial intelligence and ultrasonographers with different skills in diagnosing intussusception in children and identifying indications for surgery.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3-36 months with suspected ileocolic intussusception

Exclusion Criteria:

* Children younger than 3 months or older than 36 months with suspected ileocolic intussusception

Ages: 3 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged 3-36 months with suspected ileocolic intussusception
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-04-09 (Actual); Primary Completion 2023-05-10 (Estimated); Study Completion 2023-05-10 (Estimated)

PRIMARY OUTCOMES:
Ultrasound diagnosis of ileocolic intussusception | April 9, 2023 to May 10, 2023
  Ultrasound diagnosis of ileocolic intussusception

SECONDARY OUTCOMES:
Surgical indication of ileocolic intussusception identified by ultrasound | April 9, 2023 to May 10, 2023
  Surgical indication of ileocolic intussusception identified by ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Hongkui Yu，, Principal Investigator — Guangzhou Women and Children's Medical Center
Locations (1):
- Hongkui Yu， MD, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
For non-commercial use in research, you can contact Prof. Hongkui Yu to get the data at hongkuiyu@126.com.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: After May 20, 2023
Access Criteria: For non-commercial use in research, you can contact Prof. Hongkui Yu to get the data at hongkuiyu@126.com.